CLINICAL TRIAL: NCT06011798
Title: A Phase 2b, Prospective, Multicenter, Randomized, Double-Masked, Active-Controlled Study to Assess the Efficacy and Safety of Repeat Intravitreal Injections of Foselutoclax (UBX1325) in Patients With Diabetic Macular Edema
Brief Title: Assess the Efficacy and Safety of Repeat Intravitreal Injections of Foselutoclax (UBX1325) in Patients With DME (ASPIRE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UBX1325-04
Record Dates: First submitted 2023-08-02; First posted 2023-08-25 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Macular Edema; Retinal Disease; Macular Edema; Diabetes Mellitus; Diabetic Retinopathy; Retinal Degeneration; Retinal Diseases; Eye Diseases; Edema
Keywords: DME
MeSH Terms: conditions — Retinal Diseases; Macular Edema; Diabetes Mellitus; Diabetic Retinopathy; Retinal Degeneration; Eye Diseases; Edema | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Anti-VEGF control arm (Active Comparator): Prior to randomization, participants will receive 3 IVT injections of aflibercept over 4-week intervals. Upon randomization, participants will receive 2 mg aflibercept (50 μl of 40 μg/μl solution) IVT on Day 1, Weeks 8, and 16. A sham procedure will also be administered on Day 1.
  Interventions: Drug: Aflibercept
- foselutoclax arm (Experimental): Prior to randomization, participants will receive 3 IVT injections of aflibercept over 4-week intervals. Upon randomization, participants will receive 10 μg foselutoclax (50 μl of 0.2 μg/μl solution) IVT on Day 1 and Weeks 8 and 16. 2 mg aflibercept (50 μl of 40 μg/μl solution) will also be administered on Day 1.
  Interventions: Drug: Aflibercept; Drug: foselutoclax

INTERVENTIONS:
Drug: Aflibercept — Anti-VEGF control
Drug: foselutoclax — Experimental drug
  Other Names: UBX1325
  Arms: foselutoclax arm

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of multiple doses of foselutoclax (UBX1325) in patients with Diabetic Macular Edema. The main questions the study aims to answer are:

* Assess the efficacy of foselutoclax compared to aflibercept
* Assess the safety and tolerability of foselutoclax

DETAILED DESCRIPTION:
This study is intended to assess the efficacy and safety of foselutoclax, a phosphate pro-drug, and its active parent molecule (UBX0601, a BCL-xL inhibitor) following repeat intravitreal (IVT) injections of foselutoclax in patients with Diabetic Macular Edema (DME).

Approximately 50 patients will be enrolled and randomized 1:1 into either the foselutoclax arm,10 μg given 8 weeks apart, or the control arm of aflibercept, 2 mg every 8 weeks in order to assess the primary objective. All patients will be followed for approximately 36 weeks.

The injector will be unmasked but the evaluator will remain masked throughout the study.

This study will enroll participants ≥18 years of age with active DME disease despite treatment, with best corrected visual acuity (BCVA) between 70 to 30 Early Treatment Diabetic Retinopathy Study (ETDRS) letters (equivalent to 20/40 to 20/250 on the Snellen chart). Once patients meet inclusion/exclusion criteria, patients will receive 3 run-in injections of aflibercept approximately 4 weeks apart, with the last aflibercept injection 4-6 weeks prior to Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years.
* Patients with nonproliferative DR and DME
* Center-involved DME with Central Subfield Thickness (CST) ≥325-900 μm
* BCVA in the SE (most affected) of 70 to 30 ETDRS letters (equivalent to 20/40 to 20/250 on the Snellen chart)

Exclusion Criteria:

* Concurrent disease in the study eye (SE) or structural damage, other than DME, that could compromise BCVA, prevent BCVA improvement, require medical or surgical intervention during the study period, confound interpretation of the results, or interfere with assessment of toxicity or Color Fundus Photography (CFP) in the SE.
* Significant media opacities, including cataract, or posterior capsule opacification, which might interfere with VA, assessment of toxicity, or fundus imaging in either eye.
* Any medical condition that is uncontrolled and may prevent participation in this study, as determined by the Investigator or disqualify individuals from enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bhisitkul, MD, Ph.D., Study Director — Unity Biotechnology, Inc.
Locations (19):
- United States (19):
  - California Retina Consultants, Bakersfield, California
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Salehi Retina Institute Inc., Huntington Beach, California
  - Bay Area Retina Associates, Walnut Creek, California
  - Advanced Vision Research Institute, Longmont, Colorado
  - Rand Eye Institute, Deerfield Beach, Florida
  - Florida Eye Associates, Melbourne, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - University Retina and Macula Associates, Lemont, Illinois
  - Midwest Eye, Carmel, Indiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Sierra Eye Associates, Reno, Nevada
  - EyeHealth Northwest, Portland, Oregon
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Vision Research Solutions, PLLC, Philadelphia, Pennsylvania
  - Retina Consultants of Carolina, Greenville, South Carolina
  - Retina Research Institution of Texas, Abilene, Texas
  - Austin Retina Associates, Round Rock, Texas
  - Retina Center of Texas, Southlake, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anti-VEGF Control Arm | Foselutoclax Arm
Started | 26 | 26
Completed | 23 | 24
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-VEGF Control Arm | Foselutoclax Arm | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (8.73) | 66.2 (7.57) | 66.1 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 22 | 23 | 45
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 21 | 22 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Average of Week 20 and Week 24 in BCVA by ETDRS Letter
Description: Mean change from baseline to the average of Week 20 and Week 24 in Best-Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) letter
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: change in ETDRS letters
Arm/Group | Anti-VEGF Control Arm | Foselutoclax Arm
Number analyzed (Participants) | 26 | 26
change in ETDRS letters | 5.1 (1.35) | 3.7 (1.36)

2. Secondary Outcome: Assess Other Efficacy Outcome - Changes in BCVA From Baseline to Week 36
Description: Changes in BCVA (ETDRS letters) from baseline to Week 36
Time Frame: 36 weeks
Measure: Least Squares Mean (Standard Error); unit: change in ETDRS letters
Arm/Group | Anti-VEGF Control Arm | Foselutoclax Arm
Number analyzed (Participants) | 23 | 24
change in ETDRS letters | 4.7 (1.63) | 4.6 (1.59)

3. Secondary Outcome: Assess Other Efficacy Outcome - Changes in CST From Baseline to Week 36
Description: Change in Central Subfield Thickness (CST) as measured in microns from baseline to Week 36
Time Frame: 36 weeks
Measure: Least Squares Mean (Standard Error); unit: microns
Arm/Group | Anti-VEGF Control Arm | Foselutoclax Arm
Number analyzed (Participants) | 23 | 24
microns | 9.2 (23.69) | -1.9 (23.33)

4. Secondary Outcome: Assess Other Efficacy Outcome - Rescue Metrics
Description: At any visit, including Unscheduled visits, patients who exhibited increase in disease activity, were allowed to be rescued with aflibercept. Increase in disease activity was defined as ANY of the following:
  * Worsening CST by ≥75 µm from baseline per SD-OCT
  * A ≥10 letter decrease in BCVA compared to baseline
  * New clinically significant blood or heme present compared to previous visit
  * PI discretion (rationale to be documented in the EDC)
Time Frame: 36 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Anti-VEGF Control Arm | Foselutoclax Arm
Number analyzed (Participants) | 26 | 26
percentage of participants
  No Rescues | 61.5 | 34
  1 Rescue | 23.1 | 34.6
  > = 2 Rescues | 15.4 | 30.8

5. Secondary Outcome: Assess Safety Outcome - Safety and Tolerability
Description: Number of participants with treatment-emergent adverse event (TEAE)
Time Frame: 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-VEGF Control Arm | Foselutoclax Arm
Number analyzed (Participants) | 26 | 26
Participants
  Participants with at least one TEAE | 15 | 22
  Participants with at least one Ocular TEAE in Study Eye | 12 | 19
  Participants with at least one related Ocular TEAE in Study Eye | 8 | 8
  Participants with at least one Ocular TESAE in Study Eye | 1 | 0
  Participants with at least one Ocular TEAE in Non-Study Eye | 2 | 6
  Participants with at least one related Ocular TEAE in Non-Study Eye | 1 | 0
  Participants with at least one non-ocular TESAE | 5 | 5

6. Secondary Outcome: Ocular Safety and Tolerability
Description: Ocular Safety is evaluated by incidence of ocular Treatment Emergent Adverse Events (TEAEs).
Time Frame: 36 weeks
Population: Subjects with at least one ocular TEAE in study eye
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-VEGF Control Arm | Foselutoclax Arm
Number analyzed (Participants) | 26 | 26
Participants
  subjects with at least one ocular TEAE in study eye | 12 | 19
  diabetic retinal oedema | 8 | 15
  conjunctival haemorrhage | 8 | 15
  conjunctival hyperaemia | 22 | 2
  punctate keratitis | 2 | 1
  cataract aggravated | 10 | 1
  posterior capsule opacification | 0 | 2
  conjunctivochalasis | 0 | 1
  diabetic retinopathy | 1 | 0
  dry eye | 0 | 1
  retinal detachment | 1 | 0
  subretinal fluid | 0 | 1
  visual acuity reduced | 0 | 1
  vitreous detachment | 0 | 1
  vitreous floaters | 0 | 1
  hordeolum | 0 | 1
  corneal abrasion | 1 | 0

ADVERSE EVENTS:
Time Frame: Consent through Study Week 36, including a 12 week run-in period (for a total of 48 weeks). After the subject consented and completed all screening procedures confirming eligibility, they proceeded to the Run-in period to receive 3 injections of aflibercept 4 weeks apart.
Groups:
- Anti-VEGF Control Arm - Run-In Period; Foselutoclax Arm - Run-In Period: Prior to randomization, participants will receive 3 IVT injections of aflibercept over 4-week intervals.
Arm/Group | Anti-VEGF Control Arm - Run-In Period | Foselutoclax Arm - Run-In Period | Anti-VEGF Control Arm | Foselutoclax Arm
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 5/26 | 5/26
Other Adverse Events (participants affected / at risk) | 2/26 | 0/26 | 15/26 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-VEGF Control Arm - Run-In Period (N=26) | Foselutoclax Arm - Run-In Period (N=26) | Anti-VEGF Control Arm (N=26) | Foselutoclax Arm (N=26)
Retinal detachment (Eye disorders) | NA | NA | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | NA | NA | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | NA | NA | 0 (0) | 1 (1)
Localized Infection (Infections and infestations) | NA | NA | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | NA | NA | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | NA | NA | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | NA | NA | 1 (1) | 1 (1)
Shock hypoglycaemic (Metabolism and nutrition disorders) | NA | NA | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | NA | NA | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | NA | NA | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-VEGF Control Arm - Run-In Period (N=26) | Foselutoclax Arm - Run-In Period (N=26) | Anti-VEGF Control Arm (N=26) | Foselutoclax Arm (N=26)
Diabetic retinal oedema (Study eye) (Eye disorders) | 0 (0) | 0 (0) | 8 (8) | 15 (15)
Conjunctival haemorrhage (Study eye) (Eye disorders) | 2 (2) | 0 (0) | 4 (4) | 5 (5)
Conjunctival hyperaemia (Study eye) (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Punctate keratitis (Study eye) (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Diabetic retinal oedema (non-study eye) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Posterior capsule opacification (Study eye) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT06011798/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT06011798/SAP_001.pdf